CLINICAL TRIAL: NCT05140681
Title: Influence of Flap Position on Soft Tissue Regrowth, Keratinized Tissue Increase and Postoperative Discomfort Following Fibre Retention Osseous Resective Surgery (FibReORS): a 6-month Split-mouth RCT With Multilevel Analysis.
Brief Title: Influence of Flap Position Following FibReORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FibReORSTurin
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis; Periodontal Diseases
Keywords: periodontitis; flap position; soft tissue regrowth
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apical group (Experimental): FibReORS with apically flap positioning 2 mm below the bone crest (apical group)
  Interventions: Procedure: FibReORS with apically positioned flap (apical position)
- Crestal group (Active Comparator): FibReORS with apically flap positioning at the level of bone crest (crestal group).
  Interventions: Procedure: FibReORS with apically positioned flap (crestal position)

INTERVENTIONS:
Procedure: FibReORS with apically positioned flap (apical position) — Periodontal surgery including flap elevation. root surface scaling, bone remodeling and suture of the flap at 2 mm subcrestal position
  Arms: apical group
Procedure: FibReORS with apically positioned flap (crestal position) — Periodontal surgery including flap elevation. root surface scaling, bone remodeling and suture of the flap at either a crestal position
  Arms: Crestal group

SUMMARY:
There is lack of data in literature on keratinized tissue increase after FibReORS in relation to primary flap position. This study has been designed as a split-mouth randomized trial to assess the influence of flap position after FibReORS. 16 patients were recruited and treated. The placement of the flap 2 mm apically to the bone crest instead at the bone level would be a viable approach to increase KT width without delaying wound healing. The extent of post-operative discomfort/pain was not influenced by primary flap position.

ELIGIBILITY:
Inclusion Criteria:

1) diagnosis of severe chronic periodontitis (corresponding to grade III or IV according to the actual classification); 2) good general health; 3) full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) < 20%; 4) at least two contralateral sextants with residual PDs of > 5 mm and persisting bleeding on probing (BoP) at posterior natural teeth 3 months after the completion of cause-related therapy

Exclusion Criteria:

1) pregnancy and lactation; 2) smoking > 10 cigarettes/day; 3) intake of antibiotics in the previous 6 months. In addition, teeth with degree II or III mobility, horizontal bone loss higher than 1/3 of the root length or designed as abutment for prosthetic rehabilitation were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Amount of soft tissue re-growth after FibReORS | 6 months
  The amount of regrowth is calculated from the position of the tissue at the end of the surgery

SECONDARY OUTCOMES:
Amount of KT increase after FibReORS | 6 months
  The amount of KT increase is calculated from the position of the tissue at the end of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- C.I.R. Dental School. Università di Torino, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piccoli GM, Romano F, Giraudi M, La Bruna N, Citterio F, Mariani GM, Baima G, Aimetti M. Effect of post-surgical flap position on soft tissue regrowth and keratinized tissue increase following fibre retention osseous resective surgery: a 6-month randomized study with multilevel analysis. BMC Oral Health. 2023 Jul 10;23(1):472. doi: 10.1186/s12903-023-03144-2. PMID 37430291